CLINICAL TRIAL: NCT06350058
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Dose Escalation Study to Evalution the Safety, Tolerability of Inactivated Rotavirus Vaccine in a Population Aged 6 Weeks-49 Years Old
Brief Title: Phase I Clinical Trial of Inactivated Rotavirus Vaccine in a Population Aged 6 Weeks-49 Years Old
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202012005
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Inactivated Rotavirus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age group of 18-49 years old (Experimental): Using a dose escalation trial, divided into 2 dose groups with 25 participants in each group.
  Interventions: Biological: Inactivated rotavirus vaccine (low dose); Biological: Inactivated rotavirus vaccine (high dose); Biological: Placebo
- Age group of 1-5 years old (Experimental): Using a dose escalation trial, divided into 2 dose groups with 25 participants in each group.
  Interventions: Biological: Inactivated rotavirus vaccine (low dose); Biological: Inactivated rotavirus vaccine (high dose); Biological: Placebo
- Age group of 6-12 months old (Experimental): Using a dose escalation trial, divided into 2 dose groups with 25 participants in each group.
  In addition, a dose exploration trial was conducted, with a total of 225 subjects aged 6-12 weeks enrolled, with 100 participants in both high-dose and low-dose groups, and 25 participants in the placebo control group
  Interventions: Biological: Inactivated rotavirus vaccine (low dose); Biological: Inactivated rotavirus vaccine (high dose); Biological: Placebo

INTERVENTIONS:
Biological: Inactivated rotavirus vaccine (low dose) — The protein content of each dose is 2.5 μg. The antigen content shall not be less than 2000U, and each person shall receive one dose of 0.5ml.
Biological: Inactivated rotavirus vaccine (high dose) — The protein content of each dose is 5 μg. The antigen content shall not be less than 4000U, and each person shall receive one dose of 0.5ml.
Biological: Placebo — Aluminum hydroxide adjuvant.

SUMMARY:
The research objective is to evaluate the safety and tolerability of the inactivated rotavirus vaccine and explore its preliminary immunogenicity.

DETAILED DESCRIPTION:
This is a Phase I, single center, randomized, double-blind, placebo-controlled, dose escalation clinical trial conducted in Hebei Province, China. The purpose of this study is to evaluate the safety and tolerability of the inactivated rotavirus vaccine and explore its preliminary immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 6-12 weeks, 1-5 years old, 18-49 years old, able to provide legal identification;
* The subjects or the legal guardians of the subject have the ability to understand the research procedure, agree to participate in the study (or the legal guardian of the subject agrees to the child's participation in the study), and signs an informed consent form;
* The subjects or their legals guardian are able to participate in all planned follow-up visits;
* On the day of enrollment, the axillary body temperature was ≤ 37.0 ℃;
* Standards for certain groups of people:

Subjects aged ≥ 1 year: Laboratory test indicators (as specified in the protocol) within the normal range, or those with abnormalities but no clinical significance (evaluated by clinical doctors); Female participants of childbearing age: non pregnant, non lactating, and agreed to take effective contraceptive measures within 8 months after participating in the study.

Exclusion Criteria:

* Previously received any rotavirus vaccine;
* Previous history of acute gastroenteritis caused by rotavirus;
* Have a history of intussusception, congenital abnormalities in the digestive system, chronic diarrhea, and other diseases in the past;
* Have any history of severe allergies to vaccines or drugs in the past, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, and local allergic necrosis reaction (Arthurs reaction);
* Suffering from serious congenital malformations, developmental disorders, and genetic defects that may interfere with the progress or completion of the study (including but not limited to: Down syndrome, thalassemia, etc.);
* Diagnosed with congenital or acquired immunodeficiency, or suspected of having systemic diseases that may interfere with the conduct or completion of the study, such as tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus (HIV), syphilis infection, etc;
* Having a history or family history of convulsions, epilepsy, encephalopathy, and mental illness;
* Suffering from contraindications for intramuscular injection such as thrombocytopenia, any coagulation disorders, or receiving anticoagulant therapy;
* Recently receiving immunosuppressive therapy, such as systemic glucocorticoid therapy for more than 2 weeks continuously after birth or 6 months before vaccination, such as prednisone or similar drugs using >5mg/day (note: local and inhaled/nebulized steroids can be used);
* Any absence of spleen or splenectomy, functional absence of spleen caused by any circumstances;
* Hypertensive subjects (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg, suitable for adults);
* Three days prior to the first dose of the vaccine, there was an acute illness or a period of acute exacerbation of a chronic disease;
* Received inactivated vaccine within 7 days before enrollment and attenuated live vaccine within 14 days;
* Have received blood or blood related products or immunoglobulin (acceptable for hepatitis B immunoglobulin) within 3 months prior to enrollment;
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit;
* The researchers believe that there are any conditions in the subjects that may interfere with the evaluation of the research objectives;
* Standards for certain groups of people:

Subjects aged 6-12 weeks: single fetus gestational age<37 weeks or>42 weeks, birth weight<2.5kg or>4.0kg; multiple fetuses; abnormal birth process (difficult labor, instrumental midwifery) or a history of asphyxia and neurological damage; children with pathological jaundice.

Ages: 6 Weeks to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 375 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of AE | 0~30 day after vaccination
  The incidence of all adverse events within 0-30 days after each dose of vaccination
Incidence rate of SAE | From the first dose of vaccination to the 6 months after achieving the entire immunization process
  The incidence of all SAE from the start of the first dose of vaccination to the 6 months after achieving the entire immunization process

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Hebei Provincial Center for Disease Control and Prevention, Shijiangzhuang, Hebei, China